CLINICAL TRIAL: NCT01066650
Title: The Real-World Endeavor Resolute Versus XIENCE V Drug-Eluting SteNt Study: Head-to-head Comparison of Clinical Outcome After Implantation of Second Generation Drug-eluting Stents in a Real World Scenario
Brief Title: The Real-World Endeavor Resolute Versus XIENCE V Drug-Eluting Stent Study in Twente
Acronym: TWENTE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Foundation of Cardiovascular Research and Education Enschede (Other)
Responsible Party: Principal Investigator, prof. C. von Birgelen, Professor Clemens von Birgelen, Thorax Centrum Twente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TWENTE I; MST/Twente/001 (Registry Identifier: Dutch trial registry /Nederlands trial register NTR1256)
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Unstable Angina Pectoris; Coronary Stenosis; Coronary Restenosis
Keywords: TWENTE; randomized study; stent; coronary stent; drug-eluting stent; Zotarolimus; Everolimus; Xience V; Endeavor Resolute; head to head comparison; real world patients; target vessel failure; investigator initiated study; coronary artery disease; coronary arteries; atherosclerosis; non inferiority
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Angina, Unstable; Coronary Stenosis; Coronary Restenosis; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endeavor Resolute (Active Comparator)
  Interventions: Device: Endeavor Resolute (Biolinx-based Zotarolimus-eluting stent)
- Xience V (Active Comparator)
  Interventions: Device: Xience V (Everolimus-eluting stent)

INTERVENTIONS:
Device: Endeavor Resolute (Biolinx-based Zotarolimus-eluting stent) — Drug eluting Stent
  Other Names: Endeavor Resolute stent
  Arms: Endeavor Resolute
Device: Xience V (Everolimus-eluting stent) — Drug eluting stent
  Other Names: Xience V drug eluting stent
  Arms: Xience V

SUMMARY:
The TWENTE Study is a single center prospective single-blinded randomized study. Randomization will involve the type of Drug-Eluting Stent (DES) used in study population. Patients will be blinded to the type of DES they will receive. The general practitioner of the patient will be requested not to disclose this information to the patient. Analysts who perform the data analyses will be blinded to the type DES used as well.

DETAILED DESCRIPTION:
Primary research questions

To investigate whether the clinical outcome following the randomized implantation of the Endeavor Resolute® versus XIENCE V® drug-eluting stent is similar, as assessed in a non-inferiority setting by comparing target-vessel failure (TVF) of both stents. We want to compare for both drug-eluting stents the combined endpoint of death, myocardial infarction or revascularization related to the target-vessel, as well as death or myocardial infarction that cannot be related to a significant flow obstruction in another vessel or to another cause. According to current literature, non-inferiority of Endeavor resolute ® and XIENCE V® is expected. But the non-inferiority of Endeavor resolute and XIENCE V® is not tested in a controlled randomized trial yet.

ELIGIBILITY:
Inclusion Criteria:

* Indication for PCI with DES implantation based on VVC/ESC guidelines and/or clinical decision of interventional cardiologist
* Age ≥ 18 years and mentally capable to give an informed consent
* Signed informed consent

Exclusion Criteria:

* Patients with ST-elevation myocardial infarction (STEMI) or an ST- elevation myocardial infarction equivalent requiring primary PCI or rescue PCI
* Patients in whom the revascularization procedure is planned to be performed in a staged approach
* Renal failure requiring haemodialysis
* Patient is currently participating in an investigational drug or device study that has been not completed
* In the investigators opinion patient has a co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
* Life expectancy less than 1 year
* Patients in whom during PCI there is no indication for DES use and/or if the operator chooses not to use a DES based on the clinical situation, the patient will be excluded.
* If the choice of DES is dictated by logistic reasons e.g. the required DES dimensions is provided by one manufacturer only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1391 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
comparing target-vessel failure (TVF) of both stents | 1 year

SECONDARY OUTCOMES:
the efficacy, safety, clinical short- and long-term outcome, and the acute angiographic results of the implantation of two second-generation drug-eluting stents | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: C. von Birgelen, MD,PhD,Prof, Principal Investigator — Thorax Centrum Twente
Locations (1):
- Medisch Spectrum Twnete, Enschede, Overijssel, Netherlands

REFERENCES:
- [Derived] van Vliet D, Pinxterhuis TH, Ploumen EH, Kok MM, Buiten RA, Zocca P, Roguin A, Schotborgh CE, Anthonio RL, Danse PW, Benit E, Aminian A, Doggen CJM, von Birgelen C. Impact of diabetes on three-year outcome after coronary stenting in patients with polyvascular atherosclerotic disease - a secondary analysis of the randomized TWENTE trials. Int J Cardiol Heart Vasc. 2025 Jul 6;59:101741. doi: 10.1016/j.ijcha.2025.101741. eCollection 2025 Aug. PMID 40687396
- [Derived] Pinxterhuis TH, Ploumen EH, Doggen CJM, van Vliet D, Kok MM, Zocca P, Hartmann M, van Houwelingen KG, Stoel MG, de Man FHAF, Linssen GCM, von Birgelen C. Sex and age-specific 10-year mortality after coronary stenting: an analysis of two randomized trials. Eur Heart J Open. 2025 Jan 29;5(1):oeaf006. doi: 10.1093/ehjopen/oeaf006. eCollection 2025 Jan. PMID 39959922
- [Derived] Pinxterhuis TH, Ploumen EH, van Vliet D, Gert van Houwelingen K, Stoel MG, de Man FH, Hartmann M, Zocca P, Linssen GC, Geelkerken RH, Doggen CJ, von Birgelen C. Ten-year mortality after treating obstructive coronary atherosclerosis with contemporary stents in patients with or without concomitant peripheral arterial disease. Atherosclerosis. 2024 May;392:117488. doi: 10.1016/j.atherosclerosis.2024.117488. Epub 2024 Mar 26. PMID 38598970
- [Derived] Pinxterhuis TH, Ploumen EH, Zocca P, Doggen CJM, Schotborgh CE, Anthonio RL, Roguin A, Danse PW, Benit E, Aminian A, Hartmann M, Linssen GCM, von Birgelen C. Impact of premature coronary artery disease on adverse event risk following first percutaneous coronary intervention. Front Cardiovasc Med. 2023 Sep 7;10:1160201. doi: 10.3389/fcvm.2023.1160201. eCollection 2023. PMID 37745109
- [Derived] Pinxterhuis TH, Ploumen EH, Doggen CJM, Hartmann M, Schotborgh CE, Anthonio RL, Roguin A, Danse PW, Benit E, Aminian A, Linssen GCM, von Birgelen C. First myocardial infarction in patients with premature coronary artery disease: insights into patient characteristics and outcome after treatment with contemporary stents. Eur Heart J Acute Cardiovasc Care. 2023 Nov 16;12(11):774-781. doi: 10.1093/ehjacc/zuad098. PMID 37619976
- [Derived] Pinxterhuis TH, Ploumen EH, Zocca P, Doggen CJM, Schotborgh CE, Anthonio RL, Roguin A, Danse PW, Benit E, Aminian A, Stoel MG, Linssen GCM, Geelkerken RH, von Birgelen C. Outcome after percutaneous coronary intervention with contemporary stents in patients with concomitant peripheral arterial disease: A patient-level pooled analysis of four randomized trials. Atherosclerosis. 2022 Aug;355:52-59. doi: 10.1016/j.atherosclerosis.2022.05.002. Epub 2022 May 20. PMID 35641327
- [Derived] von Birgelen C, van der Heijden LC, Basalus MW, Kok MM, Sen H, Louwerenburg HW, van Houwelingen KG, Stoel MG, de Man FH, Linssen GC, Tandjung K, Doggen CJ, van der Palen J, Lowik MM. Five-Year Outcome After Implantation of Zotarolimus- and Everolimus-Eluting Stents in Randomized Trial Participants and Nonenrolled Eligible Patients: A Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2017 Mar 1;2(3):268-276. doi: 10.1001/jamacardio.2016.5190. PMID 28114618
- [Derived] van Houwelingen KG, Sen H, Lam MK, Tandjung K, Lowik MM, de Man FH, Louwerenburg JH, Stoel MG, Hartmann M, Linssen GC, Doggen CJ, von Birgelen C. Three-year clinical outcome after treatment of chronic total occlusions with second-generation drug-eluting stents in the TWENTE trial. Catheter Cardiovasc Interv. 2015 Feb 15;85(3):E76-82. doi: 10.1002/ccd.25713. Epub 2014 Nov 1. PMID 25339110
- [Derived] Sen H, Lam MK, Tandjung K, Lowik MM, Stoel MG, de Man FH, Louwerenburg JH, van Houwelingen GK, Linssen GC, Doggen CJ, Basalus MW, von Birgelen C. Complex patients treated with zotarolimus-eluting resolute and everolimus-eluting Xience V stents in the randomized TWENTE trial: comparison of 2-year clinical outcome. Catheter Cardiovasc Interv. 2015 Jan 1;85(1):74-81. doi: 10.1002/ccd.25464. Epub 2014 Mar 14. PMID 24585502
- [Derived] Tandjung K, Sen H, Lam MK, Basalus MWZ, Louwerenburg JHW, Stoel MG, van Houwelingen KG, de Man FHAF, Linssen GCM, Said SAM, Nienhuis MB, Lowik MM, Verhorst PMJ, van der Palen J, von Birgelen C. Clinical outcome following stringent discontinuation of dual antiplatelet therapy after 12 months in real-world patients treated with second-generation zotarolimus-eluting resolute and everolimus-eluting Xience V stents: 2-year follow-up of the randomized TWENTE trial. J Am Coll Cardiol. 2013 Jun 18;61(24):2406-2416. doi: 10.1016/j.jacc.2013.04.005. Epub 2013 Apr 16. PMID 23602769
- [Derived] Tandjung K, Basalus MW, Sen H, Stoel MG, van Houwelingen KG, Louwerenburg JH, de Man FH, Linssen GC, Said SA, Kleijne MA, van der Palen J, von Birgelen C. Women treated with second-generation zotarolimus-eluting resolute stents and everolimus-eluting xience V stents: insights from the gender-stratified, randomized, controlled TWENTE trial. Catheter Cardiovasc Interv. 2013 Sep 1;82(3):396-405. doi: 10.1002/ccd.24848. Epub 2013 Mar 8. PMID 23359390
- [Derived] Sen H, Tandjung K, Basalus MW, Lowik MM, van Houwelingen GK, Stoel MG, Louwerenburg HW, de Man FH, Linssen GC, Nijhuis R, Nienhuis MB, Verhorst PM, van der Palen J, von Birgelen C. Comparison of eligible non-enrolled patients and the randomised TWENTE trial population treated with Resolute and Xience V drug-eluting stents. EuroIntervention. 2012 Oct;8(6):664-71. doi: 10.4244/EIJV8I6A104. PMID 22581199
- [Derived] von Birgelen C, Basalus MW, Tandjung K, van Houwelingen KG, Stoel MG, Louwerenburg JH, Linssen GC, Said SA, Kleijne MA, Sen H, Lowik MM, van der Palen J, Verhorst PM, de Man FH. A randomized controlled trial in second-generation zotarolimus-eluting Resolute stents versus everolimus-eluting Xience V stents in real-world patients: the TWENTE trial. J Am Coll Cardiol. 2012 Apr 10;59(15):1350-61. doi: 10.1016/j.jacc.2012.01.008. Epub 2012 Feb 15. PMID 22341737